CLINICAL TRIAL: NCT06441786
Title: A Metacognitive Group Therapy of Depression and Anxiety in Youth With Autism: Feasibility, Acceptability and Effect in a Clinical Open Trial
Brief Title: A Metacognitive Group Therapy of Depression and Anxiety in Youth With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UUMCT001
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Depression

STUDY DESIGN:
Intervention Model Description: A clinical open trial evaluating feasibility, acceptability, as well as treatment effects measured before, after and at 6-month follow-up, for a 10-week group treatment based on metacognitive therapy, for adolescents aged 15-18 years of age with anxiety and/or depression and an autism diagnosis. The study is conducted at two psychiatric clinics for children and youth.
  The treatment structure was adjusted before the inclusion of Group 4 (Sep 2026), resulting in three individual sessions and five group sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A metacognitive group therapy of depression and anxiety in youth with autism (Experimental): A within group design where one clinical manualized intervention, Metacognitive therapy (MCT) for anxiety and depression, is offered in a 10-session group format to adolescents. The therapists have received special training in MCT and are experienced in using the methods. The treatment is delivered face-to-face.
  Interventions: Behavioral: A metacognitive group therapy of depression and anxiety in youth with autism

INTERVENTIONS:
Behavioral: A metacognitive group therapy of depression and anxiety in youth with autism — The treatment model is based on Adrian Wells' transdiagnostic A-M-C model and treatment structure described in Wells (2009) "Metacognitive therapy for anxiety and depression". The group treatment is delivered in 10 weekly sessions.

SUMMARY:
The goal of this open clinical trial is to try out and evaluate a group metacognitive treatment protocol, for adolescents aged 15-18 years of age with anxiety and/or depression and an autism diagnosis.

The main questions it aims to answer are:

1. How does the recruitment to the study work and what is the retention rate?
2. What is the level of participant compliance?
3. Is the treatment adherence satisfactory, are there any practical problems with treatment delivery?
4. Are the outcome measures and assessment procedures feasible?
5. Do the participants accept the treatment, are there any reports of adverse effects?
6. What are the preliminary effects of the treatment regarding

   1. Symptoms of anxiety and/or depression
   2. Quality of life
   3. Functional impairment
   4. Subjective level of stress
   5. Central metacognitive processes
7. Are changes in metacognitive processes related to changes in anxiety and depression?

The participants will partake in metacognitive group treatment of 10 sessions following an initial screening.

DETAILED DESCRIPTION:
Participants in the study are youth (15 to 18 years of age) seeking help for anxiety and depression within child and youth psychiatry. There will a consecutive inclusion to form 6 treatment groups with 6 persons in each. The groups will meet once every week. Assessments will take place at pre- and post-treatment as well as at 6-month follow-up. Some metacognitive processes will also be monitored at each group session. The therapists have undergone a specialist training in metacognitive therapy and are experienced in using the methods. The main focus of the study is on feasibility, acceptability and preliminary effects of the treatment. These will be analyzed with paired sample t-test on primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age of 15 to 18 years
* Seeking medical care PRIMA psychiatric clinic for children and youth in Stockholm
* Diagnoses of anxiety disorder or depression as well as autism established in a clinical interview
* Mastering the Swedish language enough to take part of the treatment
* Willingness/ability to participate after receiving information about what participation entails

Exclusion Criteria:

* Assessed to meet one of the following diagnoses: Bipolar syndrome, alcohol use syndrome, substance use syndromes, psychotic symptoms and affective syndromes with psychotic symptoms and antisocial personality disorder.
* Assessed to have a high suicide risk.
* Assessed to have extensive self-harm behavior or moderate to high risk of such.
* Participating in other psychological treatment or about to start such treatment during the time interval of the study.
* Has not had stable medication in the last month or is planning a deposit/medication adjustment during the time interval of the study.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Revised Children's Anxiety and Depression Scale (RCADS) | Change from pre intervention to treatment completion at 10 weeks and at a 6 month follow-up
  A self-report that measures symptoms of anxiety and depression.

SECONDARY OUTCOMES:
Brunnsviken Brief Quality of life questionnaire (BBQ) | Change from pre intervention to treatment completion at 10 weeks and at a 6 month follow-up
  Measure of quality of life with a total score ranging from 0 to 96 with a higher score indicating a higher quality of life. The scores of each of the six primary questions regarding perceived quality of life within an area of life are multiplied with the score of an item measuring the perceived importance of the area in question.
Metacognitions Questionnaire - 30 items version (MCQ-30) | Change from pre intervention to treatment completion at 10 weeks and at a 6 month follow-up
  A self-report measuring metacognitive assumptions and processes.
Cognitive Attentional Syndrome Scale (CAS-1) | Change from pre intervention to treatment completion at 10 weeks and at a 6 month follow-up
  A self-report measuring the presence of Cognitive Attentional Syndrome
Child Sheehan Disability Scale (CSDS) | Change from pre intervention to treatment completion at 10 weeks and at a 6 month follow-up
  A subjective appraisal of functional impairment related to familial, social and vocational aspects of life.
Perceived Stress Scale 10 (PSS-10) | Change from pre intervention to treatment completion at 10 weeks and at a 6 month follow-up.
  A questionnaire that aims to measure symptoms of stress. It contains 10 items that are scored on a range between 0 (never) to 4 (very often). The total score range is between 0-40 and a higher score reflects higher levels of perceived stress.

OTHER OUTCOMES:
Negative Effects Questionnaire, 20 items Child (NEQ 20C) | After treatment completion at 10 weeks.
  A self-report measuring negative effects of the treatment and some aspects related to acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Timo Hursti, Ph.D., Principal Investigator — Uppsala University
Locations (1):
- PRIMA Child and Youth Psychiatry, Handen, Haninge, Stockholm County, Sweden